CLINICAL TRIAL: NCT04369677
Title: Thermoregulation Among Individuals With First-episode Psychosis
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: Nicholas Breitborde (Other)
Responsible Party: Sponsor-Investigator, Nicholas Breitborde, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2020H0066
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Psychosis; First Episode Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First-Episode Psychosis: Twenty individuals with FEP will complete a 24-hour continuous assessment of core body temperature using a CorTemp ingestible sensor (HQInc., Palmetto, FL).
- Healthy: Twenty age-matched individuals with no psychotic disorder will complete a 24-hour continuous assessment of core body temperature using a CorTemp ingestible sensor (HQInc., Palmetto, FL).

SUMMARY:
The project will evaluate thermoregulatory processes among individuals with and without first-episode psychosis.

DETAILED DESCRIPTION:
The project will evaluate thermoregulatory processes among individuals with and without first-episode psychosis.

Aim 1: Assess whether individuals with first-episode psychosis have differences in mean temperature and diurnal temperature variation as compared to individuals without psychosis.

Aim 2: Examine whether mean temperature and temperature variation during periods of rest and activity are different between individuals with first-episode psychosis versus people without psychosis.

Aim 3: Explore the association between current core body temperature and current ratings of psychotic symptomatology among individuals with first-episode psychosis.

Study participants will complete baseline assessments (e.g., symptoms, functioning, and sleep) and then complete a 24-36 hour ambulatory assessment period in which core temperature, activity, sleep, and heart rate variability will be tracked continuously and symptom severity will be assessed sporadically using a symptom rating app on their smart phone. .Then they will complete a second study visit to repeat baseline assessments.

ELIGIBILITY:
Eligibility for Individuals with First-Episode Psychosis:

1. Diagnosis of a schizophrenia-spectrum disorder or mood disorder with psychotic features as determined using the Structured Clinical Interview for the DSM-5 .
2. Less than 5 years since the onset of frank psychotic symptoms as determined using the Symptom Onset in Schizophrenia Inventory.
3. No evidence of a pre-existing intellectual disability defined as a premorbid IQ >70 as estimated using the Reading subtest of the Wide Range Achievement Test-4.

Eligibility for Individuals without First-Episode Psychosis:

1. No diagnosis of a schizophrenia-spectrum disorder or mood disorder with psychotic features as determined using the Structured Clinical Interview for the DSM-5.
2. No evidence of a pre-existing intellectual disability defined as a premorbid IQ >70 as estimated using the Reading subtest of the Wide Range Achievement Test-4.

Eligibility for Individuals with and without First-Episode Psychosis:

1. Ages 18 - 35
2. No evidence of swallowing difficulties as assessed using the Swallowing Disturbance Questionnaire [SDQ]. defined as (i) a score <5 on the SDQ oral phase questions, (ii) a score <11.5 on the laryngopharygeal phase SDQ questions, and a total SDQ score < 12.5.
3. Not meeting diagnostic criteria for a substance use disorder over the past month as determined using the Structured Clinical Interview for the DSM-5 .
4. No current or past diagnosis of a medical condition known to affect thermoregulatory Functioning as assessed using the Health Conditions that Affect Thermoregulation questionnaire
5. Per recommendations from the manufacturer of the CorTemp continuous temperature sensor, we will not enroll:

   1. Individuals who weigh less than 80 pounds
   2. Individuals diagnosed with known or suspected obstructive diseases of the gastrointestinal tract
   3. Individuals with a history of gag reflex disorders or impairments
   4. Individuals with previous or scheduled gastrointestinal surgery
   5. Individuals having felinization of the esophagus
   6. Individuals with conditions that would result in hypomotility of the GI tract.
   7. Individuals scheduled to undergo Magnetic Resonance Imaging or Nuclear Magnetic Resonance in the next month
   8. Individuals with cardiac pacemaker or other implanted electric medical devices

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eligibility for Individuals with First-Episode Psychosis:
  1. Diagnosis of a schizophrenia-spectrum disorder or mood disorder with psychotic features as determined using the Structured Clinical Interview for the DSM-5 .
  2. Less than 5 years since the onset of frank psychotic symptoms as determined using the Symptom Onset in Schizophrenia Inventory.
  3. No evidence of a pre-existing intellectual disability defined as a premorbid IQ >70 as estimated using the Reading subtest of the Wide Range Achievement Test-4.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2025-04-03 (Estimated); Study Completion 2025-04-03 (Estimated)

PRIMARY OUTCOMES:
Differences in mean temperature and diurnal temperature variation | 24 hour intervals
  Differences in mean temperature and diurnal temperature variation in individuals with first-episode psychosis as compared to individuals without psychosis.
Differences in mean temperature and temperature variation during periods of rest and activity | 24 hour intervals
  Differences in mean temperature and temperature variation during periods of rest and activity between individuals with first-episode psychosis versus people without psychosis.
Association of core body temperature and ratings of psychotic symptomatology in FEP | 24 hour intervals
  Association between core body temperature and ratings of psychotic symptomatology among individuals with first-episode psychosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Harding Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu BY, Cullen CE, Eide CE, Williams CC, Apfeldorf WJ. Antidepressant-induced sweating alleviated by aripiprazole. J Clin Psychopharmacol. 2008 Dec;28(6):710-1. doi: 10.1097/JCP.0b013e31818d6b67. No abstract available. PMID 19011447
- [Background] Vybiral S, Jansky L. The role of dopaminergic pathways in thermoregulation in the rabbit. Neuropharmacology. 1989 Jan;28(1):15-20. doi: 10.1016/0028-3908(89)90061-0. PMID 2927577
- [Background] Heh CW, Herrera J, DeMet E, Potkin S, Costa J, Sramek J, Hazlett E, Buchsbaum MS. Neuroleptic-induced hypothermia associated with amelioration of psychosis in schizophrenia. Neuropsychopharmacology. 1988 May;1(2):149-56. doi: 10.1016/0893-133x(88)90006-1. PMID 3251495
- [Background] Rubinstein G. Schizophrenia, infection and temperature. An animal model for investigating their interrelationships. Schizophr Res. 1993 Aug;10(2):95-102. doi: 10.1016/0920-9964(93)90043-i. PMID 8398951
- [Background] Lkhagvasuren B, Nakamura Y, Oka T, Sudo N, Nakamura K. Social defeat stress induces hyperthermia through activation of thermoregulatory sympathetic premotor neurons in the medullary raphe region. Eur J Neurosci. 2011 Nov;34(9):1442-52. doi: 10.1111/j.1460-9568.2011.07863.x. Epub 2011 Oct 6. PMID 21978215
- [Background] Hayashida S, Oka T, Mera T, Tsuji S. Repeated social defeat stress induces chronic hyperthermia in rats. Physiol Behav. 2010 Aug 4;101(1):124-31. doi: 10.1016/j.physbeh.2010.04.027. Epub 2010 May 10. PMID 20438740
- [Background] Keeney AJ, Hogg S, Marsden CA. Alterations in core body temperature, locomotor activity, and corticosterone following acute and repeated social defeat of male NMRI mice. Physiol Behav. 2001 Sep 1-15;74(1-2):177-84. doi: 10.1016/s0031-9384(01)00541-8. PMID 11564466
- [Background] Radonjic NV, Petronijevic ND, Vuckovic SM, Prostran MS, Nesic ZI, Todorovic VR, Paunovic VR. Baseline temperature in an animal model of schizophrenia: long-term effects of perinatal phencyclidine administration. Physiol Behav. 2008 Feb 27;93(3):437-43. doi: 10.1016/j.physbeh.2007.10.003. Epub 2007 Oct 10. PMID 17996259
- [Background] Horvath G, Kekesi G, Petrovszki Z, Benedek G. Abnormal Motor Activity and Thermoregulation in a Schizophrenia Rat Model for Translational Science. PLoS One. 2015 Dec 2;10(12):e0143751. doi: 10.1371/journal.pone.0143751. eCollection 2015. PMID 26629908
- [Background] Chong TW, Castle DJ. Layer upon layer: thermoregulation in schizophrenia. Schizophr Res. 2004 Aug 1;69(2-3):149-57. doi: 10.1016/s0920-9964(03)00222-6. PMID 15469188
- [Background] Arnold VK, Rosenthal TL, Dupont RT, Hilliard D. Redundant clothing: a readily observable marker for schizophrenia in the psychiatric emergency room population. J Behav Ther Exp Psychiatry. 1993 Mar;24(1):45-7. doi: 10.1016/0005-7916(93)90007-j. PMID 8370796
- [Background] Shiloh R, Schapir L, Bar-Ziv D, Stryjer R, Konas S, Louis R, Hermesh H, Munitz H, Weizman A, Valevski A. Association between corneal temperature and mental status of treatment-resistant schizophrenia inpatients. Eur Neuropsychopharmacol. 2009 Sep;19(9):654-8. doi: 10.1016/j.euroneuro.2009.04.010. Epub 2009 Jun 2. PMID 19493658
- [Background] Mazerolle SM, Ganio MS, Casa DJ, Vingren J, Klau J. Is oral temperature an accurate measurement of deep body temperature? A systematic review. J Athl Train. 2011 Sep-Oct;46(5):566-73. doi: 10.4085/1062-6050-46.5.566. PMID 22488144
- [Background] Palmier-Claus JE, Ainsworth J, Machin M, Barrowclough C, Dunn G, Barkus E, Rogers A, Wykes T, Kapur S, Buchan I, Salter E, Lewis SW. The feasibility and validity of ambulatory self-report of psychotic symptoms using a smartphone software application. BMC Psychiatry. 2012 Oct 17;12:172. doi: 10.1186/1471-244X-12-172. PMID 23075387
- [Background] First, M.B., et al., Structured Clinical Interview for DSM-5-Research Version2015, Arlington, VA: American Psychiatric Association.
- [Background] Perkins DO, Leserman J, Jarskog LF, Graham K, Kazmer J, Lieberman JA. Characterizing and dating the onset of symptoms in psychotic illness: the Symptom Onset in Schizophrenia (SOS) inventory. Schizophr Res. 2000 Jul 7;44(1):1-10. doi: 10.1016/s0920-9964(99)00161-9. PMID 10867307
- [Background] Wilkinson, G.S. and G.J. Robertson, Wide Range Achievement Test (WRAT4)2006, Lutz, FL: PAR, Inc
- [Background] Manor Y, Giladi N, Cohen A, Fliss DM, Cohen JT. Validation of a swallowing disturbance questionnaire for detecting dysphagia in patients with Parkinson's disease. Mov Disord. 2007 Oct 15;22(13):1917-21. doi: 10.1002/mds.21625. PMID 17588237
- [Background] Cohen JT, Manor Y. Swallowing disturbance questionnaire for detecting dysphagia. Laryngoscope. 2011 Jul;121(7):1383-7. doi: 10.1002/lary.21839. Epub 2011 Jun 10. PMID 21671239
- [Background] Cheshire WP Jr. Thermoregulatory disorders and illness related to heat and cold stress. Auton Neurosci. 2016 Apr;196:91-104. doi: 10.1016/j.autneu.2016.01.001. Epub 2016 Jan 6. PMID 26794588
- [Background] Auther, A., C. Smith, and B. Cornblatt, Global Functioning: Social Scale (GF: Social). Glen Oaks, NY: Zucker-Hillside Hospital, 2006.
- [Background] Niendam, T., et al., Global Functioning: Role Scale (GF: Role). Los Angeles, CA: University of California, Los Angeles, 2006.
- [Background] Hays, R.D., S. Prince-Embury, and H.Y. Chen, RAND-36 Health Status Inventory1998, San Antonio, TX: The Psychological Corporation.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518